CLINICAL TRIAL: NCT03017885
Title: An Active Surveillance to Monitor the Real World Safety in Indian Patients Prescribed Nintedanib for the Treatment of Locally Advanced, Metastatic or Locally Recurrent Non Small Cell Lung Cancer (NSCLC) of Adenocarcinoma Tumor Histology After First Line Chemotherapy
Brief Title: Post Marketing Surveillance of Nintedanib in Indian Patients With Non-small Cell Lung Cancer (NSCLC) After First-line Therapy
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0272
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Patients who started treatment with nintedanib & docetaxel after 23rd January, 2017 and have discontinued the drug at the time of participation in the active surveillance.
- Group B: Patients who started treatment with nintedanib & docetaxel after 23rd January, 2017 and are continuing the drug at the time of participation in the active surveillance .
- Group C: Patients who have been newly prescribed nintedanib & docetaxel at the time of participation in the active surveillance.

SUMMARY:
This active surveillance aims to collect the safety data of 100 NSCLC patients treated with nintedanib per the approved Indian label within 2 years from the date of commercial availability of the drug in India (23rd January 2017). The objective is to look at the safety of nintedanib in the real world setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with locally advanced and/or metastatic NSCLC of stage IIIB or IV, or recurrent NSCLC and adenocarcinoma histology after first line chemotherapy who have initiated or will initiate nintedanib & docetaxel according to the package insert after the commercial availability of drug in India (23rd January 2017).
* Patients in whom it is possible to obtain voluntary informed consent from either the patient or patient's legally authorised representative (applicable for Group B and C patients).
* Patients in whom data collection is possible from the medical records (applicable for Group A and B patients).
* Further inclusion criteria apply.

Exclusion Criteria:

* Patients who were previously treated with nintedanib.
* Patients who are positive for endothelial growth factor receptor (EGFR) mutations or anaplastic lymphoma kinase (ALK) rearrangements
* Patients who are participating in a clinical trial.
* Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This active surveillance aims to collect the safety data of 100 NSCLC patients treated with nintedanib per the approved Indian label within 2 years from the date of commercial availability of the drug in India (23rd January 2017).
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2022-09-24 (Actual); Study Completion 2022-09-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- India (11):
  - Zydus Hospitals and Healthcare Research Pvt. Ltd, Anand
  - Narayana Hrudyalaya, Bangalore
  - Manipal Hospitals, Bengaluru
  - HCG Hospital, Bengaluru
  - Sparsh Hospitals and Critical Care, Bhubaneshwar
  - Action Cancer Hospital, Delhi, Delhi
  - Apollo Health City Hospital, Hyderabad
  - Yashoda Hospitals, Hyderabad
  - Chittaranjan National Cancer Institute, Kolkata
  - Rajiv Gandhi Cancer Institute and Research Centre, New Delhi
  - SRM Institute of Medical Science, Vadapalani

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An active surveillance to monitor the real-world safety in Indian patients prescribed nintedanib as per approved Indian Label for the treatment of locally advanced, metastatic or recurrent non-small cell lung cancer (NSCLC) of adenocarcinoma tumour histology after first-line chemotherapy.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Nintedanib and Docetaxel: Group A: Group A: Non-small cell lung cancer (NSCLC) patients who had started treatment with the approved Indian labels of nintedanib and docetaxel after 23rd January 2017 and had discontinued the drug at the time of participation in the active surveillance.
- Nintedanib and Docetaxel: Group B: Group B: Non-small cell lung cancer (NSCLC) patients who started treatment with the approved Indian labels of nintedanib and docetaxel after 23rd January 2017 and were continuing the drug at the time of participation in the active surveillance.
- Nintedanib and Docetaxel: Group C: Group C: Non-small cell lung cancer (NSCLC) patients were newly prescribed the approved Indian labels nintedanib and docetaxel at the time of participation in the active surveillance.
- Single Agent Docetaxel: Group I: Group I: Non-small cell lung cancer (NSCLC) patients who started treatment with docetaxel after 23rd January 2017 and had discontinued the drug at the time of participation in the active surveillance. Patients who received the single agent docetaxel were not followed up after the baseline visit as per the study design.
- Single Agent Docetaxel: Group II: Group II: Non-small cell lung cancer (NSCLC) patients who had started treatment with docetaxel after 23rd January 2017 and were continuing the drug at the time of participation in the active surveillance. Patients who received the single agent docetaxel were not followed up after the baseline visit as per the study design.
- Single Agent Docetaxel: Group III: Group III: Non-small cell lung cancer (NSCLC) patients who were newly prescribed docetaxel at the time of participation in the active surveillance. Patients who received the single agent docetaxel were not followed up after the baseline visit as per the study design.
Period: Overall Study
Arm/Group | Nintedanib and Docetaxel: Group A | Nintedanib and Docetaxel: Group B | Nintedanib and Docetaxel: Group C | Single Agent Docetaxel: Group I | Single Agent Docetaxel: Group II | Single Agent Docetaxel: Group III
Started | 9 | 5 | 9 | 1 | 3 | 1
Completed (Completed treatment) | 0 | 0 | 0 | 1 (Completed is actually not applicable (NA). As per protocol, Patients who received the single agent docetaxel were not followed up after the baseline visit as per the study design.) | 3 (Completed is actually not applicable (NA). As per protocol, Patients who received the single agent docetaxel were not followed up after the baseline visit as per the study design.) | 1 (Completed is actually not applicable (NA). As per protocol, Patients who received the single agent docetaxel were not followed up after the baseline visit as per the study design.)
Not Completed | 9 | 5 | 9 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Progression of disease | 4 | 3 | 4 | 0 | 0 | 0
Not completed — Other than listed | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 3 | 0 | 0 | 0
Not completed — Change to other anti-cancer therapy | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Entered set (ES): Included patients who signed the Informed Consent Form (ICF) and met the eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib and Docetaxel: Group A | Nintedanib and Docetaxel: Group B | Nintedanib and Docetaxel: Group C | Single Agent Docetaxel: Group I | Single Agent Docetaxel: Group II | Single Agent Docetaxel: Group III | Total
Number analyzed (Participants) | 9 | 5 | 9 | 1 | 3 | 1 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.7 (5.8) | 59.8 (9.2) | 57.0 (12.1) | 39.0 (NA) — For single count, Standard Deviation can not be calculated. | 61.7 (11.9) | 56.0 (NA) — For single count, Standard Deviation can not be calculated. | 58.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 0 | 1 | 0 | 7
  Male | 7 | 2 | 8 | 1 | 2 | 1 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence of All Adverse Drug Reactions (ADRs) in Nintedanib and Docetaxel Treated Patients
Description: Incidence of all Adverse drug reactions (ADRs) in nintedanib and docetaxel treated patients.
  An Adverse Event (AE) was considered as an Adverse drug reaction (ADR) if either the physician who reported the AE or the sponsor assessed its causal relationship as 'related'.
  The incidence rate were calculated using number of patients with respective events divided by time at risk expressed as [100 pt -yrs].
Time Frame: From first drug administration until 28 days after the last drug administration, up to 586 days.
Population: Only patients who were treated with nintedanib and docetaxel and were included in the treated set (TS).
  TS: all patients who signed the informed consent form (ICF), met the eligibility criteria and had take at least one dose of study medication.
  Results are reported for overall nintedanib and doxetaxel group. According to the protcol, it was not planned to compare all 3 groups of nintedanib and docetaxel.
Measure: Number (95% Confidence Interval); unit: Patients per 100 patient years
Groups:
- Nintedanib and Docetaxel: Non-small cell lung cancer (NSCLC) patients who had started treatment with the approved Indian labels of nintedanib and docetaxel (all Groups).
Arm/Group | Nintedanib and Docetaxel
Number analyzed (Participants) | 23
Patients per 100 patient years | 17.9 [2.2 to 64.7]

2. Primary Outcome: Incidence Rate of All Serious Adverse Events (SAEs) in Nintedanib and Docetaxel Treated Patients
Description: Incidence rate of all Serious Adverse Events (SAEs) in nintedanib and docetaxel treated patients.
  All Adverse Events (AEs) that occurred between the first intake of nintedanib plus docetaxel and within 28 days (inclusive) after the last intake were considered 'treatment emergent'.
  The incidence rate were calculated using number of patients with respective events divided by time at risk expressed as [100 pt -yrs].
Time Frame: From first drug administration until 28 days after the last drug administration, up to 586 days.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Patients per 100 patient years
Arm/Group | Nintedanib and Docetaxel
Number analyzed (Participants) | 23
Patients per 100 patient years | 25.3 [12.7 to 45.4]

3. Secondary Outcome: Percentage of Patients Who Required Nintedanib Dose Reductions
Description: Percentage of patients who required nintedanib dose reductions.
Time Frame: From first drug administration until 28 days after the last drug administration, up to 586 days.
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Nintedanib and Docetaxel
Number analyzed (Participants) | 23
Percentage of Participants | 4.3

4. Secondary Outcome: Number of Patients Who Discontinued Study Drug Permanently Due to Adverse Events
Description: Number of patients who discontinued study drug permanently due to adverse events.
Time Frame: From first drug administration until last drug administration, up to 558 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib and Docetaxel
Number analyzed (Participants) | 23
Participants | 2

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after the last drug administration, up to 586 days. All-cause mortality: Up to 51.5 months after first drug administration.
Description: As defined in protocol safety data was not collected for patients treated with single agent docetaxel as they were not followed up after the baseline visit.
  There was no plan to compare all 3 nintedanib and docetaxel groups according to the protocol.
  Only patients who were treated with nintedanib and docetaxel and were included in the treated set (TS).
  TS: all patients who signed the informed consent form (ICF), met the eligibility criteria and had take at least one dose of study medication.
Groups:
- Docetaxel and Nintedanib: Non-small cell lung cancer (NSCLC) patients who had started treatment with the approved Indian labels of nintedanib and docetaxel (all Groups).
Arm/Group | Docetaxel and Nintedanib
All-Cause Mortality (participants affected / at risk) | 9/23
Serious Adverse Events (participants affected / at risk) | 9/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel and Nintedanib (N=23)
Gastroenteritis (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Loss of consciousness (Nervous system disorders) | 1
Unresponsive to stimuli (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
Study enrolled lower number of patients than the planned sample size due to low recruitment at the selected sites. The study was real-world active surveillance hence no examinations were mandated. Information collected as per clinical practice was available which may not have been consistent across patients and study duration.

The extent of retrospectively collected study data for patients in Group A and I were dependent on the information available in medical records at the time of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review Prior to any Submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI´s intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT03017885/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT03017885/SAP_001.pdf